CLINICAL TRIAL: NCT00003012
Title: A Prospective Randomized Comparison of CMF Versus Sequential Epirubicin Followed by SMF as Adjuvant Chemotherapy for Women With Early Breast Cancer
Brief Title: Combination Chemotherapy Following Surgery in Treating Women With Early Stage Breast Cancer
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Scottish Cancer Therapy Network (Other)
Organization: National Cancer Institute (NCI) (NIH)
Allocation: Randomized | Purpose: Treatment
Other Study IDs: CDR0000065590; SCTN-BR9601; EU-97013
Record Dates: First submitted 1999-11-01; First posted 2004-04-06 (Estimated); Last update posted 2013-11-06 (Estimated); Status verified 2008-11

CONDITIONS: Breast Cancer
Keywords: stage II breast cancer; stage IIIA breast cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — CMF regimen; Cyclophosphamide; Epirubicin; Fluorouracil; Methotrexate

INTERVENTIONS:
Drug: CMF regimen
Drug: cyclophosphamide
Drug: epirubicin hydrochloride
Drug: fluorouracil
Drug: methotrexate

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die. It is not yet known which combination chemotherapy regimen is more effective following surgery for breast cancer.

PURPOSE: Randomized phase III trial to study the effectiveness of combination chemotherapy consisting of cyclophosphamide, methotrexate, and fluorouracil with or without epirubicin in treating women who have early stage breast cancer.

DETAILED DESCRIPTION:
OBJECTIVES: I. Compare the effects of 4 courses of epirubicin followed by 4 courses of cyclophosphamide/methotrexate/fluorouracil (CMF) versus 8 courses of CMF as adjuvant chemotherapy in women with node positive early breast cancer, as measured by overall and event free survival from the date or randomization. II. Compare the effects of 4 courses of epirubicin followed by 4 courses of CMF with 8 courses of CMF as adjuvant chemotherapy in these patients, as measured by acute and chronic toxicities. III. Compare the effects of 4 courses of epirubicin followed by 4 courses of CMF versus 8 courses of CMF as adjuvant chemotherapy in these patients, as measured by quality of life.

OUTLINE: This is a randomized, multicenter study. Patients are randomized into 2 treatment arms within 4 weeks of surgery. Treatment begins within 6 weeks of surgery. One treatment arm receives 8 courses of cyclophosphamide/methotrexate/fluorouracil (CMF) given intravenously (IV) every 3 weeks. The other arm receives 4 courses of epirubicin followed by 4 courses of CMF given IV every 3 weeks. Patients are followed annually for 10 years.

PROJECTED ACCRUAL: A total of 1,000 patients will be accrued over 3 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS: Histologically confirmed, early stage, unilateral invasive breast cancer of TNM stages T0 - T3, N0-1, M0, i.e., Histologically proven axillary node metastases OR Lymph node negative Not locally advanced If supraclavicular node is enlarged or suspicious of metastasis, negative biopsy for supraclavicular node metastases required No evidence of any other metastases clinically or on routine staging investigations No past history of pure in situ carcinoma in either breast Primary tumor is completely excised

PATIENT CHARACTERISTICS: Age: Not specified Sex: Female Performance status: Not specified Hematopoietic: Neutrophil count greater than 2,000/mm3 Platelet count greater than 100,000/mm3 No evidence of sepsis Hepatic: Adequate hepatic function Bilirubin normal AST/ALT normal Renal: Adequate renal function Creatinine less than 1.2 mg/dL Cardiovascular: No clinically significant cardiovascular disease Other: No prior or concurrent other malignancy except adequately treated basal or squamous cell carcinoma of the skin or in situ carcinoma of the cervix Not pregnant or nursing Fertile patients must use effective contraception

PRIOR CONCURRENT THERAPY: Biologic therapy: Not specified Chemotherapy: No prior chemotherapy Endocrine therapy: Prior tamoxifen allowed Radiotherapy: No prior radiotherapy Surgery: See Disease Characteristics

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 1000 (Estimated)
Dates: Start 1996-10

CONTACTS AND LOCATIONS:
Overall Officials: Chris Twelves, MD, BMedSci, FRCP, Study Chair — University of Glasgow
Locations (10):
- United Kingdom (10):
  - University Hospitals of Leicester, Leicester, England
  - Aberdeen Royal Infirmary, Aberdeen, Scotland
  - Ninewells Hospital and Medical School, Dundee, Scotland
  - Western General Hospital, Edinburgh, Scotland
  - Beatson Oncology Centre, Glasgow, Scotland
  - University of Glasgow, Glasgow, Scotland
  - Raigmore Hospital, Inverness, Scotland
  - Royal Alexandra Hospital, Paisley, Scotland
  - Ayr Hospital, Ayr
  - Falkirk Royal Infirmary, Falkirk

REFERENCES:
- [Background] Earl H, Hiller L, Dunn JA, et al.: The National Epirubicin Adjuvant Trial (NEAT) and Scottish Cancer Trials Breast Group (SCTBG) br9601 randomized phase III adjuvant early breast cancer trials: the updated definitive joint analysis. [Abstract] J Clin Oncol 25 (Suppl 18): A-534, 11s, 2007.
- [Background] Poole CJ, Earl HM, Hiller L, Dunn JA, Bathers S, Grieve RJ, Spooner DA, Agrawal RK, Fernando IN, Brunt AM, O'Reilly SM, Crawford SM, Rea DW, Simmonds P, Mansi JL, Stanley A, Harvey P, McAdam K, Foster L, Leonard RC, Twelves CJ; NEAT Investigators and the SCTBG. Epirubicin and cyclophosphamide, methotrexate, and fluorouracil as adjuvant therapy for early breast cancer. N Engl J Med. 2006 Nov 2;355(18):1851-62. doi: 10.1056/NEJMoa052084. PMID 17079759
- [Background] Poole CJ, Earl HM, Dunn JA, et al.: NEAT (National Epirubicin Adjuvant Trial) and SCTBG BR9601 (Scottish Cancer Trials Breast Group) phase III adjuvant breast trials show a significant relapse-free and overall survival advantage for sequential ECMF. [Abstract] Proceedings of the American Society of Clinical Oncology 22: A-13, 4, 2003.
- [Result] Bartlett JM, Munro A, Cameron DA, Thomas J, Prescott R, Twelves CJ. Type 1 receptor tyrosine kinase profiles identify patients with enhanced benefit from anthracyclines in the BR9601 adjuvant breast cancer chemotherapy trial. J Clin Oncol. 2008 Nov 1;26(31):5027-35. doi: 10.1200/JCO.2007.14.6597. Epub 2008 Sep 2. PMID 18768436
- [Derived] Braunstein M, Liao L, Lyttle N, Lobo N, Taylor KJ, Krzyzanowski PM, Kalatskaya I, Yao CQ, Stein LD, Boutros PC, Twelves CJ, Marcellus R, Bartlett JM, Spears M. Downregulation of histone H2A and H2B pathways is associated with anthracycline sensitivity in breast cancer. Breast Cancer Res. 2016 Feb 6;18(1):16. doi: 10.1186/s13058-016-0676-6. PMID 26852132